CLINICAL TRIAL: NCT01691365
Title: Oxidative Damage and Inflammation in Obese Diabetic Emirati Subjects Supplemented With Antioxidants and B-vitamins: a Randomized Placebo-controlled Trail
Brief Title: Effects of Antioxidants and B Vitamins Supplements on Inflammation in Obese Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Collaborators: Tawam Hospital (Other)
Responsible Party: Principal Investigator, Salah Gariballa, Professor, United Arab Emirates University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMHS
Record Dates: First submitted 2012-09-11; First posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes; Obesity
Keywords: Antioxidant; vitamins; Diet
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Vitamins; Antioxidants; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamins pills (Active Comparator): antioxidant and B vitamins vitamins vitamin
  --------------------------------------------------------------------------------
  Interventions: Dietary Supplement: vitamins
- pills (Placebo Comparator): MICROCRYSTALLINE CELLULOSE
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: vitamins — a capsule of antioxidant vitamins 221mg of alpha tocopherol and 167mg of vitamin C and B-group vitamins (1.67 mg folic acid, 1.67mg vitamin B-2, 20 mg vitamin B-6, 0.134 mg vitamin B-12) or an identical placebo daily for 90 days
  Other Names: Antioxidants; B vitamins
  Arms: vitamins pills
Drug: Placebo — Placebo Capsule shell (Hydroxypropylmethyl cellulose, Hydroxypropylcellulose, Propylene glycol as stabilizer, Colour-Titanium dioxide)
  Arms: pills

SUMMARY:
Substantial evidence shows that diets incorporating antioxidants and B-group vitamins can offer significant protection against infections and cardiovascular disease (CVD) especially in diabetic patients. The proposed study will determine whether improvements in antioxidants and B-group vitamins in diabetic patients who are known to have a high risk of CVD will lead to a clinical benefit

DETAILED DESCRIPTION:
Following informed written consent 96 diabetic patients will be randomly assigned to receive either an oral dose of daily B-group vitamins (5 mg folic acid, 5mg vitamin B-2, 50 mg vitamin B-6, 0.4 mg vitamin B-12) and antioxidant vitamins [800 IU (727mg) of a-tocopherol and 500mg of vitamin C] [n=48], or no supplements [n= 48] daily for 90 days. All subjects will have three assessments, at baseline, 3, and 12 months post-randomisation. The assessment will include markers of inflammation, endothelial dysfunction, oxidative stress, antioxidants, total plasma homocysteine and risk of infections. A fasting 15-ml of blood will be taken for measurements of total plasma homocysteine concentration, markers of inflammation, endothelial dysfunction, oxidative damage and vitamin concentrations. Further information on clinical variables which may influence endothelial dysfunction, antioxidant capacity, immunity and diabetes control status will be collected and adjusted for during analysis.

Potential Significance- the study will help to clarify the temporal relationships between , markers of inflammation, endothelial dysfunction and oxidative stress and risk of infections and form the basis of appropriate intervention strategies to minimise the long-term complications associated with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes mellitus

Exclusion Criteria:

* severe chronic clinical or psychiatric disease,
* participating in other intervention trials,
* on dietary supplements and
* those unable to give an informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Inflammation | 3 months
Oxidative damage | 3 months

SECONDARY OUTCOMES:
Antioxidant status | 3 months

OTHER OUTCOMES:
Infections | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Salah Gariballa, MD, Principal Investigator — United Arab Emirates University

REFERENCES:
- [Derived] Gariballa S, Alkaabi J, Yasin J, Al Essa A. Total adiponectin in overweight and obese subjects and its response to visceral fat loss. BMC Endocr Disord. 2019 Jun 3;19(1):55. doi: 10.1186/s12902-019-0386-z. PMID 31159801